CLINICAL TRIAL: NCT03693014
Title: A Phase II Trial of Hypofractionated Radiotherapy in Patients With Limited Progression on Immune Checkpoint Blockade
Brief Title: A Study of Several Radiation Doses for Patients With Progression on Immunotherapy/Checkpoint Inhibitors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-359
Record Dates: First submitted 2018-10-01; First posted 2018-10-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Cancer; Melanoma Cancer; Lung Cancer; Bladder Cancer; Renal Cancer; Head/Neck Cancers
Keywords: Radiation; Immunotherapy/Checkpoint Inhibitors; 18-359
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms | interventions — Radiosurgery; Ipilimumab; Nivolumab; pembrolizumab; atezolizumab

STUDY DESIGN:
Intervention Model Description: This is an open label Phase 2 screening trial in subjects.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic Body Radiotherapy (Experimental): Image Guided, Stereotactic Body Radiotherapy (27 Gy over 3 fractions) to 1-3 lesions. Treatment with the checkpoint inhibitor will continue until progression at the discretion of the treating physician or unacceptable toxicity.
  Interventions: Radiation: Stereotactic Body Radiotherapy; Biological: Ipilimumab, Nivolumab, Pembrolizumab or Atezolizumab

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — (27 Gy over 3 fractions)
Biological: Ipilimumab, Nivolumab, Pembrolizumab or Atezolizumab — The checkpoint inhibitor that the patient was already receiving should be continued according to the standard schedule and dose of administration as determined by the treating physician. Immune Checkpoint Inhibitors include Ipilimumab (Melanoma) Nivolumab (Melanoma, Renal, NSCLC), Pembrolizumab (Melanoma, NSCLC), Atezolizumab (Bladder)

SUMMARY:
Drugs called checkpoint inhibitors help the immune system fight cancer. When the effectiveness of these drugs wears off, it may be possible to renew their effectiveness by combining it with a special type of radiation therapy called stereotactic body radiation therapy (SBRT). SBRT is a commonly used type of radiation therapy that gives high dose radiation with high precision to tumors in 1-5 treatments. Radiation therapy, such as SBRT can also treat sites of metastases. The use of checkpoint inhibitors in combination with SBRT has been suggested to improve the immune response against cancer but has not been tested in a formal clinical trial. Up to three lesions can be treated with SBRT. This study only allows checkpoint inhibitors that are already approved by the Federal Drug Agency (FDA) for the treatment of your disease. All radiation therapy will be done on machines which are FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated an IRB approved written informed consent form in accordance with regulatory and institutional guidelines.
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study obligations.
* Males and females ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Histologically confirmed metastatic cancer of any histology for which there is an FDA indication for an immune checkpoint inhibitor including melanoma, lung, bladder, renal and head/neck cancers.
* Patient has been receiving treatment with an immune checkpoint inhibitor including but not limited to ipilimumab, nivolumab, avelumab, durvalumab, pembrolizumab, atezolizumab, and tremelimumab for at least 2 months. A combination of these therapies is also permitted. No max prior lines of therapy.
* Patient has evidence of limited progression (up to 5 lesions either new or increase in at least 25% in the cross-sectional diameter of a known lesion) on most recent systemic imaging as determined by the treating physician. Patients with greater than 5 lesions can be included after discussion with the study investigators.
* Patient must be eligible to continue to receive an immune checkpoint inhibitor after radiotherapy.
* Subjects must have at least two lesions:

  * One lesion must be safely amenable to irradiation in the opinion of the treating radiation oncologist. This can be a lesion that was previously irradiated if it is deemed appropriate by the treating physician and principal investigator. Standard MSKCC re-irradiation dose constraints must be met.
  * At least one, not-to-be-irradiated lesion measurable by CT or MRI per RECIST 1.1 criteria.
* Prior palliative or curative radiotherapy must be completed at least 14 days prior to treatment.
* Immunosuppressive doses of systemic medication, such as steroids or absorbed topical steroids (doses >10mg/day prednisone or equivalent) must be discontinued at least 14 days prior to radiotherapy administration.
* Women of childbearing potential must have a negative serum within 7 days prior to treatment, or urine pregnancy test (within 24 hours) (minimum sensitivity 25 IU/L or equivalent units of HCG). Women of childbearing potential must agree to follow instructions for method(s) of contraception from time of enrollment for the duration of treatment.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year.

Notes:

* Women who are not of childbearing potential i.e., who are postmenopausal or surgically sterile as well as azoospermia men do not require contraception.
* Azoospermic males, and women of childbearing potential who are continuously not heterosexually active, are exempt from contraceptive requirements. However, they still must have a pregnancy test.
* Exclusion Criteria:

  * Active brain metastases (untreated brain metastases or growth on imaging as defined below) or leptomeningeal disease are not allowed. Subjects with brain metastases are eligible if these have been treated and there is no MRI (or CT if MRI contraindicated) evidence of progression for at least 8 weeks after treatment for these metastases is complete and within 28 days prior to first study treatment.
  * Any medical disorder that, in the opinion of the investigator, might increase the risk associated with study participation or interferes with the interpretation of study results.
  * Prior active malignancy within the previous 3 years except for locally curable cancers such as basal or squamous skin cancer, superficial bladder, low risk prostate cancer, breast, or cervix cancer. If other prior malignancy was active within prior 3 years, enrollment requires approval of a principal investigator.
  * Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
  * Subjects requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents for greater than 5 days) or other immunosuppressive medications within 14 days of study drug administration should be excluded. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * Treatment with any other chemotherapy, radiation therapy, biologics for cancer, or investigational therapy concurrently or within 14 days of enrollment
  * History of allergy to checkpoint inhibitors
  * History of severe hypersensitivity reaction to any monoclonal antibody.
  * Women must not be breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
evaluate overall response rate (ORR) | 24 weeks
  in non-irradiated lesions during the first 24 weeks after treatment initiation as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in patients with limited progression receiving hypofractionated radiotherapy. ORR rate is defined as the number of patients treated to a given arm with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Hartford Healthcare, Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm